CLINICAL TRIAL: NCT02871219
Title: A Phase II Study of Obinutuzumab and Lenalidomide in Previously Untreated Subjects With Follicular Lymphoma
Brief Title: Obinutuzumab and Lenalidomide in Treating Patients With Previously Untreated Stage II-IV Grade 1-3a Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0464; NCI-2016-01506 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0464 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Ann Arbor Stage II Grade 1 Follicular Lymphoma; Ann Arbor Stage II Grade 2 Follicular Lymphoma; Ann Arbor Stage III Grade 1 Follicular Lymphoma; Ann Arbor Stage III Grade 2 Follicular Lymphoma; Ann Arbor Stage IV Grade 1 Follicular Lymphoma; Ann Arbor Stage IV Grade 2 Follicular Lymphoma; Bulky Disease; Fatigue; Fever; Grade 3a Follicular Lymphoma; Night Sweats; Splenomegaly; Weight Loss
MeSH Terms: conditions — Fatigue; Fever; Splenomegaly; Weight Loss | interventions — Lenalidomide; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (obinutuzumab, lenalidomide) (Experimental): Patients receive obinutuzumab IV over 4-6 hours on days 1, 8, and 15 of course 1 and day 1 of cycles 2-6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, and 30. Treatment repeats every 28 days for up to 30 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR or CRu may receive up to an additional 12 cycles of lenalidomide.
  Interventions: Drug: Lenalidomide; Biological: Obinutuzumab

INTERVENTIONS:
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759

SUMMARY:
This phase II trial studies how well obinutuzumab and lenalidomide work in treating patients with previously untreated stage II-IV grade 1-3a follicular lymphoma. Immunotherapy with obinutuzumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving obinutuzumab and lenalidomide may work better in treating patients with previously untreated follicular lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of obinutuzumab combined with lenalidomide in patients with previously untreated follicular lymphoma (FL) (determined by progression-free survival [PFS] at 2 years).

SECONDARY OBJECTIVES:

I. To evaluate the safety of obinutuzumab in combination with lenalidomide in patients with untreated follicular lymphoma.

II. To evaluate the efficacy of obinutuzumab in combination with lenalidomide in subjects with follicular lymphoma as assessed by complete remission (CR) at 30 months, overall response rate (ORR), duration of response (DOR), event free survival (EFS), and overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To evaluate prognostic and predictive biomarkers relative to treatment outcomes.

OUTLINE:

Patients receive obinutuzumab intravenously (IV) over 4-6 hours on days 1, 8, and 15 of course 1 and day 1 of courses 2-6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, and 30. Treatment repeats every 28 days for up to 30 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive lenalidomide orally (PO) on days 1-21. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR or complete remission unconfirmed (CRu) may receive up to an additional 12 courses of lenalidomide.

After completion of study treatment, patients are followed up every 6 months for 18 months and then every year for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of follicular lymphoma (grades 1, 2, or 3a), untreated
* Able and willing to provide written informed consent and to comply with the study protocol
* Bi-dimensionally measurable disease, with at least one mass lesion >= 2 cm in longest diameter by computed tomography (CT), positron emission tomography (PET)/CT, and/or magnetic resonance imaging (MRI)
* Must be in need of therapy as evidenced by at least one of the following criteria:

  * Bulky disease defined as:

    * A nodal or extranodal (except spleen) mass > 7 cm in its greater diameter or,
    * At least 3 nodal or extranodal sites >= 3 cm in diameter
  * Presence of at least one B symptom:

    * Fever (> 38 C) not due to infectious etiology
    * Night sweats
    * Weight loss > 10% in the past 6 months
  * Fatigue due to lymphoma
  * Splenomegaly (> 13 cm)
  * Compression syndrome (ureteral, orbital, gastrointestinal)
  * Any of the following cytopenias due to lymphoma:

    * Hemoglobin =< 10 g/dL
    * Platelets =< 100 x 10^9/L
    * Absolute neutrophil count (ANC) < 1.5 x 10^9/L
  * Pleural or peritoneal effusion
  * Lactate dehydrogenase (LDH) > upper limit of normal (ULN) or beta-2 microglobulin > ULN
* Stage II, III, or IV disease
* Eastern cooperative oncology group (ECOG) performance status =< 2
* Absolute neutrophil count (ANC) > 1.0 x 10^9/L
* Platelet count > 75 x 10^9/L
* Serum aspartate transaminase (AST) or alanine transaminase (ALT) < 3 x upper limit of normal (ULN)
* Creatinine clearance > 30 ml/min calculated by modified Cockcroft-Gault formula
* Bilirubin < 1.5 x ULN unless bilirubin is due to Gilbert's syndrome, documented liver involvement with lymphoma, or of non-hepatic origin, in which case bilirubin should not exceed 3 g/dL
* Women of childbearing potential and men who are sexually active must practice reliable contraceptive measures started at least 4 weeks before study therapy and continued for at least 4 weeks following discontinuation therapy; females of childbearing potential must either completely abstain from heterosexual sexual contact or must use 2 methods of reliable contraception; reliable contraceptive methods include 1 highly effective method (intrauterine device, birth control pills, hormonal patches, injections, vaginal rings, or implants) and at least 1 additional method (condom, diaphragm, or cervical cap) every time they have sex with a male; males who are sexually active must be practicing complete abstinence or agree to a condom during sexual contact with a pregnant female or female of child bearing potential; men must agree to not donate sperm during and after the study
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at screening; women who are pregnant or breastfeeding are ineligible for this study; females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategies (REMS) program
* All study participants must be registered into the mandatory Revlimid REMS program, and be willing and able to comply with the requirements of the REMS program
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study

Exclusion Criteria:

* Known active central nervous system lymphoma or leptomeningeal disease
* Follicular lymphoma with evidence of diffuse large B-cell transformation
* Grade 3b follicular lymphoma
* Any prior history of other malignancy besides follicular lymphoma, unless the patient has been free of disease for >= 5 years and felt to be at low risk for recurrence by the treating physician, except:

  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of lenalidomide capsules, or put the study outcomes at undue risk
* Known history of human immunodeficiency virus (HIV), active hepatitis C virus, active hepatitis B virus infection, or any uncontrolled active systemic infection

  * Patients with inactive hepatitis B infection must adhere to hepatitis B reactivation prophylaxis unless contraindicated
* Prior use of lenalidomide
* Concurrent systemic immunosuppressant therapy (e.g., cyclosporine, tacrolimus, etc., or chronic administration glucocorticoid equivalent of > 10 mg/day of prednisone) within 28 days of the first dose of study drug
* Known anaphylaxis or IgE-mediated hypersensitivity to murine proteins or to any component of rituximab
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block, type II AV block, or 3rd degree block
* Vaccinated with live, attenuated vaccines within 4 weeks of study entry
* Lactating or pregnant subjects
* Administration of any investigational agent within 28 days of first dose of study drug
* Patients who have undergone major surgery within 14 days
* Patients with the following:

  * Bleeding diathesis or patients in whom prophylactic antithrombotic therapy is otherwise contraindicated
  * Patients with prior deep vein thrombosis (DVT), pulmonary embolism (PE), or arterial thromboembolism
  * Patients with ischemic stroke or transient ischemic attack (TIA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loretta J Nastoupil, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Akkad N, Feng L, Westin JR, Hagemeister FB, Lee HJ, Fayad L, Ahmed S, Nair R, Rodriguez MA, Strati P, Chihara D, Flowers CR, Claret L, Ibanez K, Wang M, Fowler NH, Henderson J, Davis RE, Neelapu SS, Green M, Nastoupil LJ. A phase 2 study of obinutuzumab combined with lenalidomide in previously untreated high tumor burden follicular lymphoma. Blood Adv. 2025 Sep 9;9(17):4396-4404. doi: 10.1182/bloodadvances.2025016483. PMID 40517417
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Patients receive obinutuzumab IV over 4-6 hours on days 1, 8, and 15 of course 1 and day 1 of cycles 2-6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, and 30. Treatment repeats every 28 days for up to 30 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive lenalidomide PO on days 1-21. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR or CRu may receive up to an additional 12 cycles of lenalidomide.
  Lenalidomide: Given PO
  Obinutuzumab: Given IV
Period: Overall Study
Arm/Group | Single Arm
Started | 90
Completed | 58
Not Completed | 32
Not completed — Adverse Event | 15
Not completed — Death | 3
Not completed — Progression | 3
Not completed — Infections | 7
Not completed — Infusion Related | 4

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 81
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 70
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Will be calculated and corresponding 95% confidence interval (CI) will be derived.
Time Frame: approximately 71 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm
Number analyzed (Participants) | 90
months | 70.7 [65.8 to 76.1]

2. Secondary Outcome: Complete Response
Description: The number and percentage of subjects will be tabulated.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 90
percentage of participants | 96.6 [90.4 to 99.3]

3. Secondary Outcome: Overall Response Rate (CR + Partial Response [PR])
Description: The number and percentage of subjects will be tabulated.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 90
percentage of participants | 97.70 [92.0 to 99.7]

4. Secondary Outcome: Duration of Response
Description: Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI.
Time Frame: From the time by which measurement criteria for CR or PR, whichever is recorded first, is met until death or the first date by which progressive disease is documented, assessed up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 90
percentage of participants | NA [NA to NA] — The DOR was not reached

5. Secondary Outcome: Event Free Survival
Description: Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI.
Time Frame: From the date of course 1, day 1 to the date of first documented progression, transformation to diffuse large B-cell lymphoma, initiation of new anti-lymphoma treatment, or death, assessed up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 90
percentage of participants | NA [NA to NA] — The EFS was not reached

6. Secondary Outcome: Overall Survival
Description: Kaplan-Meier methodology will be used to estimate event-free curves, median, and 95% CI.
Time Frame: From the date of course 1, day 1 to the date of death regardless of cause, assessed up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 90
percentage of participants | NA [NA to NA] — The OS was not reached

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed for up to 24 months. All-Cause Mortality monitored/assessed up to 3 years.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 3/90
Serious Adverse Events (participants affected / at risk) | 55/90
Other Adverse Events (participants affected / at risk) | 87/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Single Arm (N=90)
Blood and lymphatic systmem disorders-Other (Blood and lymphatic system disorders) | 2
Colitis (General disorders) | 3
Colonic hemorrhage (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 31
Diarrhea (Gastrointestinal disorders) | 55
Eye disorders-Other (Basal cell carcinoma (left eye rim) (Nervous system disorders) | 1
Fatigue (Nervous system disorders) | 43
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Fever (Nervous system disorders) | 21
Headache (Nervous system disorders) | 20
Hypercalcemia (Pain in extremity and hypercalcemia) (Vascular disorders) | 2
Hyperuricemia (Renal and urinary disorders) | 4
Hypotension (Vascular disorders) | 1
Infections and infestations-Other (Infections and infestations) | 2
Investigations-Other (Investigations) | 12
Investigation and-Other (Diverticulitis) (Investigations) | 1
Lung Infection (Pneumonia) (Respiratory, thoracic and mediastinal disorders) | 7
Neutrophil count decreased (Blood and lymphatic system disorders) | 19
Paroxysmal atrial tachcardia (Vascular disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10/48
Respiratory, thoracic and mediastinal disorders- Other (Pulmonary Embolims) (Respiratory, thoracic and mediastinal disorders) | 1/1
Salivary gland infection (Infections and infestations) | 1/1
Sick sinus syndrome (Respiratory, thoracic and mediastinal disorders) | 1/1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1/4
Syncope (Vascular disorders) | 2/2
Treatment related secondary malignancy (Bladder Cancer) (Renal and urinary disorders) | 2/2
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1/22
Urinary tract infection (Renal and urinary disorders) | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=90)
Abdominal Pain (Gastrointestinal disorders) | 8
Agitation (Nervous system disorders) | 1
Alanine aminotransferase increased (Renal and urinary disorders) | 3
Alkaline phosphatase increased (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 16
Anemia (Blood and lymphatic system disorders) | 7
Anorexia (Gastrointestinal disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Renal and urinary disorders) | 2
Atelectasis (Blood and lymphatic system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bloating (Gastrointestinal disorders) | 4
Blood and lymphatic system disorders-Other (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Blood and lymphatic system disorders) | 1
Blurred Vision (Nervous system disorders) | 9
Bronchial Infection (Respiratory, thoracic and mediastinal disorders) | 2
Chest pain-cardiac (Respiratory, thoracic and mediastinal disorders) | 1
Chills (Musculoskeletal and connective tissue disorders) | 6
Concentration impairment (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 44
Cough (Respiratory, thoracic and mediastinal disorders) | 28
Creatinine Increased (Blood and lymphatic system disorders) | 2
Depression (Nervous system disorders) | 2
Diarrhea (Gastrointestinal disorders) | 53
Dizziness (Nervous system disorders) | 13
Drye Eye (General disorders) | 8
Dry mouth (General disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 9
Dysgeusia (Nervous system disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23
Ear Pain (General disorders) | 1
EdemaFace (General disorders) | 2
Edema limbs (General disorders) | 14
Eye disorders-Other (Nervous system disorders) | 3
Fatigue (Nervous system disorders) | 43
Fever (General disorders) | 20
Flu like symptoms (General disorders) | 1
Flushing (Renal and urinary disorders) | 2
General disorders and administration site condtions-Other (General disorders) | 4
Headache (Nervous system disorders) | 19
Headache and Hypotension (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Renal and urinary disorders) | 2
Hypokalemia (Nervous system disorders) | 2
Infections and infestations- Other (Infections and infestations) | 1
Infusion related reaction (General disorders) | 4
Insomnia (Nervous system disorders) | 8
Investigations-Other (Nervous system disorders) | 9
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 4
Lymphedema (Infections and infestations) | 10
Lymphocyte count decreased (Blood and lymphatic system disorders) | 4
Memory Impairment (Nervous system disorders) | 10
Metabolism and nutrition disorders-Other (Metabolism and nutrition disorders) | 2
Mucositis oral (Investigations) | 3
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 41
Nasal Congestion (Blood and lymphatic system disorders) | 5
Nausea (Gastrointestinal disorders) | 27
Nervous system disorders-Other (Nervous system disorders) | 2
Neutrophil count decreased (Blood and lymphatic system disorders) | 3
Non-cardiac chest pain (Gastrointestinal disorders) | 3
Palpitations (Cardiac disorders) | 2
Papulopustular rash (Skin and subcutaneous tissue disorders) | 2
Paresthesia (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 5
Platelet count decreased (Blood and lymphatic system disorders) | 1
Portal vein thrombosis (Vascular disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8
Psychiatric disorders-Other (Nervous system disorders) | 1
Pulmonary edema (Cardiac disorders) | 1
Pulmonary fibrosis (Cardiac disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 38
Respiratory, thoracic and mediastinal disorders-Other (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis infective (Respiratory, thoracic and mediastinal disorders) | 1
Sinus bradycardia (Cardiac disorders) | 6
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 3
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 6
Skin infection (Skin and subcutaneous tissue disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 1
Thromboembolic event (Respiratory, thoracic and mediastinal disorders) | 3
Tinnitus (General disorders) | 1
Tremor (Nervous system disorders) | 4
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 21
Urinary tract infection (Renal and urinary disorders) | 4
Ventricular arrhythmia (Vascular disorders) | 1
Ventricular tachycardia (Vascular disorders) | 1
Vomiting (General disorders) | 5
Weight loss (General disorders) | 1
White blood cell decreased (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT02871219/Prot_SAP_000.pdf